CLINICAL TRIAL: NCT07109934
Title: Compare the Effect of Incentive Spirometry Versus Chest Mobilization on Oxygenation and Chest Expansion for Patient Undergoing Upper Abdominal Surgery: A Randomized Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marwa karim jabr (Other)
Collaborators: University of Baghdad (Other)
Responsible Party: Sponsor-Investigator, Marwa karim jabr, instructor, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BaghdadU
Record Dates: First submitted 2025-07-23; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Upper Abdominal Surgery
Keywords: upper abdominal surgery; Incentive spirometry; Deep breathing; Chest expansion

STUDY DESIGN:
Intervention Model Description: The sample will be chosen from the patients undergoing upper abdominal surgery at the Hospital using a simple random selection procedure. The technique of simple random sampling is extensively employed in quantitative research using survey instruments. The viability of simple random sampling in homogeneous and uniformly selected groups is demonstrated. This selection strategy ensures that all individuals have an equal chance to participate in the study, with the selection procedure being completely determined by chance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- deep breathing exercises, chest mobilization: (Experimental): The first group received a breathing exercise 2 hours after the surgery while they were completely conscious. The patients were instructed to engage in deep and gentle inspired breathing, maintain it for 3 seconds, and then exhale gently via the mouth while seated in a semi-sitting posture. During expiration, the patients were instructed to cough twice with maximum efficiency (patients were instructed to maintain a cushion in the incision area during coughing). Thereafter, the patient was provided with an incentive spirometer to be utilized 5 to 10 times daily at intervals of 2 hours. The chest mobilization was conducted five times each set, with three sets assigned to each session Individual participants independently performed chest mobilization under the guidance of a physiotherapist for the first time. The chest mobilization technique involves pulling the arms upwards to their maximum extent while inhaling appropriately during arm movement.
  Interventions: Device: deep breathing exercises, chest mobilization:
- 2. deep breathing exercises, incentive spirometry: the second group was received usual routine hospi (No Intervention)

INTERVENTIONS:
Device: deep breathing exercises, chest mobilization: — The patients were instructed to engage in deep and gentle inspired breathing, maintain it for 3 seconds, and then exhale gently via the mouth while seated in a semi-sitting posture. During expiration, the patients were instructed to cough twice with maximum efficiency (patients were instructed to maintain a cushion in the incision area during coughing). Thereafter, the patient was provided with an incentive spirometer to be utilized 5 to 10 times daily at intervals of 2 hours. The chest mobilization was conducted five times each set, with three sets assigned to each session Individual participants independently performed chest mobilization under the guidance of a physiotherapist for the first time. The chest mobilization technique involves pulling the arms upwards to their maximum extent while inhaling appropriately during arm movement.
  Arms: deep breathing exercises, chest mobilization:

SUMMARY:
This study compares the effects of incentive spirometry and chest mobilization on oxygenation and chest expansion in patients after upper abdominal surgery. It is a randomized clinical trial that aims to determine which intervention more effectively improves respiratory function. The findings likely reveal that both methods positively impact lung expansion and oxygenation, but one may be superior in enhancing recovery and preventing postoperative pulmonary complications.

DETAILED DESCRIPTION:
The most prevalent and severe type of conditions identified after upper abdomen procedures are postoperative respiratory issues. The probability of experiencing postoperative pulmonary problems increases as the incision being made during an operation approaches the diaphragm. Upper abdominal surgical operations are associated with a 20% occurrence of postoperative pulmonary problems, while lower abdominal surgeries have a lower prevalence ranging from 2% to 8%. Percutaneous upper abdomen procedures trigger a sequence of pathological reactions that may result in postoperative pulmonary problems in older individuals. Pathological responses encompass a decline in central nervous system activity, reduced mobility of the diaphragm, impaired function of the mucociliary system, decreased effectiveness of coughing, alterations in the ventilation-perfusion ratio, increased respiratory rate, and decreased pulmonary volumes and capacities.

An incentive spirometer (IS) is a feedback device designed to motivate patients to inhale deeply and generate a prolonged maximum inspiration in order to primarily open and stabilize portions of the lung affected by atelectasis. It offers mild resistance exercise yet minimizing the risk of fatigue to the diaphragm muscle.

In the context of physical activity aimed at enhancing chest expansion and ventilation, chest mobilization method is a component. It is executed by raising the arms to their maximum extent while inhaling deliberately. The chest mobilization technique facilitates the opening of individual rib cages in the upper, middle, and lower regions of the chest wall. It also enhances the mobility of the stern costal and costovertebral joints, therefore positively impacting chest movement and ventilation .

Importance of the study Recovery following surgery may be impeded by a range of symptoms including physical discomfort, psychological distress, emotional instability, and pain. Under general anesthesia during surgery, the lungs of a patient are unable to achieve complete ventilation. The discomfort resulting from the abdominal incision hinders inhalation, therefore limiting lung expansion. Postoperative pulmonary complications (PPCs) may arise, particularly when surgery is conducted in the upper abdomen region.

Individuals suffering from chronic pain disorders may experience compromised deep breathing mechanisms. This group of patients is susceptible to respiratory impairment caused by a range of factors including pneumonia, atelectasis, bronchiectasis, sleep apnea, chronic obstructive lung disease, and restrictive lung disease. Furthermore, those who have inadequate nutritional condition, excessive salivation, aspiration, gastric reflux, compromised airway clearance caused by muscle weakness or incoordination, and insufficient pulmonary reserve are more susceptible to respiratory insufficiency, morbidity, and death.

Perioperative pulmonary complications (PPCs) are frequently seen after pulmonary surgery and are linked to the duration of hospitalization, illness, death, and healthcare expenses in the public health system. Reports have indicated that the occurrence of PPCs ranges from less than 1% to 23% in major surgical procedures. About 11.5% of the occurrence of PPCs was observed in individuals who had thoracic and abdominal procedures.

Moreover, following pulmonary surgery resulted in a decrease in lung volume, diffusing capacity, and exercise capacity. The forced expiratory volume in 1 second (FEV1) is the primary indicator of co-morbidity and postoperative problems following surgery. The reduction in FEV1 following pulmonary surgery is directly linked to the disparity in lung volume resection.

Pulmonary complications can be reduced via the optimi- zation of pulmonary function, intensive pulmonary hygiene, and early ambulation.

1 Chest physiotherapy plays an impor- tant role in the treatment of atelectasis and preventing its progression to more signiﬁcant pulmonary complications following major surgeries. Pulmonary complications can be reduced via the optimi- zation of pulmonary function, intensive pulmonary hygiene, and early ambulation.

1 Chest physiotherapy plays an impor- tant role in the treatment of atelectasis and preventing its progression to more signiﬁcant pulmonary complications following major surgeries. Pulmonary complications can be reduced via the optimi- zation of pulmonary function, intensive pulmonary hygiene, and early ambulation.

1 Chest physiotherapy plays an impor- tant role in the treatment of atelectasis and preventing its progression to more signiﬁcant pulmonary complications following major surgeries. By optimizing pulmonary function, practicing rigorous pulmonary hygiene, and initiating early ambulation, it is possible to minimize pulmonary problems. The significance of chest physiotherapy is crucial in the management of atelectasis and in preventing its advancement to more severe pulmonary problems after major surgical procedures.

Respiratory and chest wall physiotherapy have been employed as preventive measures against atelectasis. Hospitalization-based respiratory exercises have demonstrated improvements in respiratory muscle strength, oxygenation, coughing mechanism, chest wall mobility, lung ventilation, as well as reduction in respiratory effort and prevention of postoperative pulmonary problems.

Prophylactic and/or postoperative physiotherapy has been extensively employed to prevent surgical complications and improve the recuperation of these individuals. Nevertheless, there is significant variation in the details of the suggested physiotherapy programs and the time of their execution (before to and/or following surgery).

Post-operative patients and those with neuromuscular or chest wall illness frequently experience atelectasis. Given that atelectasis in certain patients seems to result from frequent shallow inhalations, taking deeper breaths may be beneficial. In controlled experiments, incentive spirometers have been shown to promote lung expansion to the greatest extent possible above spontaneous breathing.

In post-surgery wards, incentive spirometry is employed to prevent and treat respiratory problems by measurement of frequent maximal inspiratory effort. This technique facilitates deep breathing and prolonged inspiration, therefore resulting in collateral ventilation. It is an objectives-driven feedback mechanism.

Historically, the primary objective of physiotherapy for lung surgery patients was to enhance chest expansion, facilitate bronchial clearing, correct posture, and improve shoulder range of motion. Recent advancements in lung volume reduction and lung transplant procedures, along with several new studies on physiotherapy in COPD patients, have introduced a fresh viewpoint to the physiotherapy approach in pulmonary surgical candidates.

The incentive spirometry (IS) is a mechanical breathing device that has been implemented in clinical medical practice. Incentive spirometry prompts the patient to take extended, deliberate deep breaths that imitate natural sighing, while also offering a visual affirmative reinforcement. Available incentive spirometers are designed to measure either the volume of inspiration (volume-oriented) or the flow rate (flow-oriented).

Diaphragmatic breathing exercises are employed to enhance the downward movement of the diaphragm during inhalation and the upward movement of the diaphragm during expiration. The advantageous outcomes of diaphragmatic breathing include alveolar inflation, mitigation of postoperative hypoxemia, enhancement of ventilation and oxygenation, reduction of respiratory effort, and augmentation of diaphragm excursion.

Postoperative pulmonary problems and arterial oxygenation preservation following laparoscopic colorectal surgery may be reduced by perioperative breathing training.

Manifestations include impaired ventilator mechanics, reduced lung compliance, and heightened respiratory effort. The much diminished lung capacities directly lead to compromised gas exchange. Multiple investigations have consistently shown arterial hypoxemia and reduced diffusion capacity during the initial postoperative phase.

The incidence of surgical complications rises with advancing age, obesity, smoking, and pre-existing lung disorders. Further variables, including the surgical site, duration of anesthesia, and post-operative risk factors such as emergency operations, insufficient preoperative education, immobilization, analgesics, and cation, have been documented to contribute to an elevated risk.

Pulmonary problems constitute the primary cause of postoperative morbidity and mortality, impacting 25-50% of patients after major abdominal surgery [3]. Moreover, these consequences can result in heightened patient suffering, elevated utilization of resources, and extended duration of hospitalization, therefore leading to a general elevation in healthcare expenses.

Operative units commonly use chest physical therapy as a means of reducing pulmonary problems. Nevertheless, the available evidence regarding its effectiveness and the trials that compare various physical rehabilitation methods are somewhat scarce. The objective of postoperative physical therapy is to enhance maximal inspiration in order to encourage the expansion of collapsed alveoli and prevent more atelectasis.

One physical therapy approach employed to address chest problems is chest resistance exercise, which involves applying resistance to the sternal and coastal regions to promote the correct alignment of respiratory muscles with respiratory rhythm. By comparison, chest expansion exercise is a comprehensive form of physical activity that combines dynamic motions of the trunk and limbs with deep breathing. This particular form of exercise has the potential to improve mobility in the chest and intercostal spaces, as well as reduce stiffness in connective tissue.

Evaluation of thoracic mobility and chest expansion is crucial for investigating causes of compromised pulmonary function, dyspnea, and reduced exercise tolerance in patients with various pulmonary or rheumatic disorders, following thoracic surgery or rib cage trauma.

Sorou, Khalil, and Sharaan, El Geneidy (2019) they conducted a study Effect of Deep Breathing Exercises versus Incentive Spirometry on Pulmonary Complications among Geriatric Patients Undergoing Upper Abdominal Surgery in Egypt, they recommended that Comparative studies which focus on comparing the effectiveness of combination of deep breathing exercises and incentive spirometer versus using each one alone, is needed to be established in gerontological nursing research.

Chaudhary, Shukla, Sairker (2023) they conducted a study an observational study on effect of breathing exercise on quality of recovery among postoperative patients in India, they state that Despite the widespread use of deep breathing exercises in patient care, there is a lack of scientific evidence supporting their effectiveness.

Although numerous studies have investigated the effect of chest physiotherapy in abdominal and thoracic surgery patients, only one publication to our knowledge has ad- dressed this topic in surgery.

the previous study has not investigated the chest mobilization technique for increasing chest expansion, oxygenation in patients undergoing upper abdominal surgery. Therefore, the purposes of the current study are to investigate the effect of combined chest mobilization with physical therapy treatment on chest expansion and oxygenation in patients undergoing upper abdominal surgery and to examine the effect of the combined chest mobilization with physical therapy treatment on the functional capacity.

There are no known published research studies on Compare the effect of deep breathing exercises with incentive spirometry chest mobilization on oxygenation and chest expansion upper abdominal surgery.

Objective(s) of the study:

1. To assess the effect of deep breathing exercises, incentive spirometry, and chest mobilization on oxygenation and chest expansion for patient undergoing upper abdominal surgery.
2. To Compare the effect of deep breathing exercises, incentive spirometry, and chest mobilization on oxygenation and chest expansion for patient undergoing upper abdominal surgery.

Research questions or hypothesis:

Is there are different between oxygenation, chest expansion for patient with upper abd surgery whom receive deep breathing and incentive spirometer combined with chest mobilization and those whom receive deep breathing and incentive spirometer?

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 18> 60 years
2. posted for upper abdominal surgery.
3. Accepted to participate in the study

Exclusion Criteria:

1. . Patients exhibiting unstable hemodynamic parameters characterized by arterial pressure below 100 mmHg systolic and below 60 mmHg diastolic, and mean arterial pressure (MAP) below 80 mmHg.
2. Surgical patients experiencing postoperative problems needing mechanical ventilation.
3. Uncooperative patients or individuals with limited comprehension or inability to proficiently operate the gadget .

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-02-22 (Estimated); Study Completion 2026-04-22 (Estimated)

PRIMARY OUTCOMES:
Tape measuring | 6 time point at which the measurement is assessed for both study and control groups divided in to tow days, 3 times per day as following after 1 hours , after 8 hours and after 16 hours
  • Tape measuring is extensively employed in to assess chest expansion, participants are directed to complete a maximal inhale and exhale, as it is a straightforward and easily detectable movement of the chest. The extent of chest expansion is determined by subtracting the thoracic circumference at the conclusion of forced inspiration from the thoracic circumference at the conclusion of forced expiration
Physiological Evaluation: | 6 time point at which the measurement is assessed for both study and control groups divided in to tow days, 3 times per day as following after 1 hours , after 8 hours and after 16 hours
  - Pulse oximetry, sometimes known as the fifth vital sign, is a rapid and non-invasive monitoring method that measures the oxygen saturation in the blood by directing visible light at particular wavelengths through tissue, typically the fingernail bed. This pulse oximeter comprises a peripheral probe and a microprocessor unit that presents a waveform, the computed oxygen saturation percentage, and the average pulse rate. Available alarms are triggered by a low SpO2 level or a pulse rate that is either tachycardia or bradycardic.

CONTACTS AND LOCATIONS:
Locations (1):
- AL-Kindi teaching hospital, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No